CLINICAL TRIAL: NCT04839757
Title: Preparing for the Use of a Dengue Vaccine in the French Caribbean Islands of Martinique and Guadeloupe : the DengueSEA Study
Brief Title: Dengue Vaccine Strategy in Children Aged 9 to 17 Years in the French Caribbean
Acronym: DengueSEA
Status: Recruiting | Type: Observational
Sponsor: University Hospital Center of Martinique (Other)
Collaborators: Ecole des Hautes Etudes en Santé Publique (Other); University Hospital Center of Guadeloupe (Unknown); Observatoire Regional de la Sante Provence-Alpes-Côte d'Azur (Other); Modélisation Mathématique des Maladies Infectieuses UMR 2000, Institut Pasteur (Unknown); Institut de Recherche en Santé Publique, France (Other); Aix Marseille Université (Other)
Responsible Party: Sponsor
Other Study IDs: 19_RIPH3_19; 2019-A02114-53 (Other: Numéro ID RCB _ ANSM)
Record Dates: First submitted 2021-03-29; First posted 2021-04-09 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Dengue; Vaccination; Seroprevalence; Infectious Disease
Keywords: dengue; seroprevalence; children; adolescents; vaccination strategy; French Carribean
MeSH Terms: conditions — Dengue; Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Dengue fever, an arbovirus transmitted by the Aedes mosquito, is a public health problem in all tropical and subtropical regions of the world. There is currently no antiviral treatment and vector control has shown its limits. The 2018 European marketing authorization of the tetravalent chimeric yellow fever / dengue vaccine (Dengvaxia®) is a major step forward in the fight against the disease. Dengvaxia® is indicated for the prevention of dengue due to serotypes DENV 1-4 in subjects aged 9 to 45 years with a history of infection with the dengue virus and living in endemic areas (seroprevalence of at least 70% in the target population).

Dengue seroprevalence data in the French Caribbean territories of Martinique and Guadeloupe dates back to 2011 and concerns only adult blood donors aged 18 to 70 years. To date, no data exists for individuals aged 9 to 17 years in the region.

In order to implement an optimal vaccine introduction strategy for these territories, the main aim of the DengueSEA study is to estimate the seroprevalence of the Dengue viruses (DENV 1-4) in 9-17 year olds giving a blood sample as part of care in hospital departments of the French Caribbean islands of Martinique and Guadeloupe.

DETAILED DESCRIPTION:
The Dengvaxia® vaccine is being implemented in a difficult context: complex administration of the vaccine with the need to perform a biological test beforehand and to administer 3 vaccine doses, inconsistent efficacy, controversies and legal actions against the manufacturer in some countries where the vaccine has been used in children under 9 years of age, and general mistrust of vaccines, particularly the most recent ones.

In Martinique and Guadeloupe, where dengue circulates in an endo-epidemic mode, outbreaks involving all four DENV serotypes were observed in 1997, 2001, 2005, 2007, 2010 and 2013. Dengue seroprevalence for the region, estimated in 18-70 year old adult blood donors in 2011, was 93.5% (95% CI [91.5-95.1]). It was 86.7% (95% CI [69.3-96.2]) in 18- to 19-year-olds. A single dengue virus infection (primary dengue) was observed in 3% of dengue-positive donors. The remainder had been infected with two or more dengue viruses. To date, no such seroprevalence data exists for individuals aged 9 to 17 years in these regions, hence the DengueSEA study.

At the same time, a survey on the acceptability of dengue vaccination, conducted among parents/legal guardians of participating children/adolescents will allow the assessment of the degree of vaccine hesitancy, particularly for Dengvaxia®, and to identify its main determinants.

In addition, Martinique and Guadeloupe were affected in 2016 by an epidemic of the Zika virus infection, which affected 50 to 60% of the population. The antigenic relationship between dengue and Zika viruses can be the cause of serological cross-reactions and could have an impact on the efficacy and tolerance of dengue vaccines in individuals with a history of Zika virus infection. This justifies the conduct of a joint seroprevalence study of Zika and dengue virus infections in the study population.

The DengueSEA study is a key towards the implementation of an optimal dengue vaccination strategy for children aged 9 to 17 years in the French Caribbean. The results of this research will also permit better organization of health care services and better management of medical resources, particularly in anticipation of future dengue epidemics in the region. Potential vaccine acceptability challenges will also be better anticipated. Finally, the constitution of a biological collection will allow the evaluation of future serological tests developed to select eligible individuals for dengue vaccination, notably with Dengvaxia®, and to carry out further seroprevalence studies on arboviruses.

ELIGIBILITY:
CHILDREN

Inclusion Criteria for children:

* Any child aged 9 to 17 years presenting to one of the hospital departments participating in the study at the University Hospitals of Martinique or Guadeloupe
* Need to take a blood sample or place a peripheral venous line for the management of the child
* Residence in Martinique or Guadeloupe since at least one year
* Information on the study given to the child and his/her parent or legal guardian
* Collection of the parent's or legal guardian's non-objection to the child's participation

Exclusion Criteria for children:

* Presence of fever or suspected acute infection
* Presence of an immune deficiency or any other dysimmune condition

PARENTS

Parental inclusion criteria ("vaccine acceptability" survey)

* Collection of the parent's or legal guardian's non-objection to participate in the Dengvaxia® vaccine acceptability survey
* Comprehension of spoken and written French

Non-inclusion criteria for parents (vaccine acceptability survey)

- None of the above

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Any child aged 9 to 17 years presenting to one of the hospital departments participating in the study at the University Hospitals of Martinique or Guadeloupe who Need to take a blood sample or place a peripheral venous line for the management of the child
  Collection of the parent's or legal guardian's non-objection to participate in the Dengvaxia® vaccine acceptability survey
Sampling Method: Probability Sample
Enrollment: 590 (Estimated)
Dates: Start 2021-06-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Dengue seroprevalence in the study population | through study completion, an average of 1 year
  Number of anti-DENV IgG positive cases, with seroneutralization in favor of previous DENV infection, divided by the total number of 9-17 year odl children/adolescents included in the DengueSEA study

SECONDARY OUTCOMES:
Frequency of primary dengue fever | through study completion, an average of 1 year
  Serum neutralisation with antibody titration by DENV serotype (DENV 1 to 4)
Temporal variation of the risk of dengue infection | through study completion, an average of 1 year
  Implementation of a mathematical prediction model, based on a dynamic mode of infection during dengue epidemics in the French Caribbean, and taking into account dengue seroprevalence and surveillance data in the region since 2001 (Public Health France, sentinel physicians network)
Seroprevalence of Zika infection | through study completion, an average of 1 year
  anti-ZIKV IgG positivity and seroneutralization in favor of a previous Zika virus infection divided by the total number of children included in the DengueSEA study
Assessment of Dengue vaccine acceptability/characterization of intentions and attitudes | through study completion, an average of 1 year
  Questionnaire developed using the "3C" model developed by the WHO SAGE group to predict the degree of vaccine hesitancy, i.e., the refusal or postponement of certain vaccinations despite the availability of these products. The factors favored by this model are confidence in the safety of the vaccine (Confidence), perception of the importance of the targeted vaccination (Complacency), and perceived difficulties in obtaining this vaccination (Convenience).

CONTACTS AND LOCATIONS:
Overall Officials: Andre CABIE, Principal Investigator — Martinique University Hospital Center
Locations (1):
- Martinique University Hospital Center, Fort-de-France, Martinique